CLINICAL TRIAL: NCT05126316
Title: Multiple-dose Safety, Pharmacokinetic and Pharmacodynamic Trial, in Subjects With Allergic Rhinitis
Brief Title: A Trial to Learn More About Repeated Monthly Injections of Lu AG09222 in Participants With Allergies to Grass Pollen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19424A
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lu AG09222 Low Dose (Experimental): Participants will receive Lu AG09222 injection at a low dose level 3 times with 4 weeks between each administration.
  Interventions: Drug: Lu AG09222
- Lu AG09222 High Dose (Experimental): Participants will receive Lu AG09222 injection at a high dose level 3 times with 4 weeks between each administration.
  Interventions: Drug: Lu AG09222
- Placebo (Placebo Comparator): Participants will receive placebo matching to Lu AG09222 injection 3 times with 4 weeks between each administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AG09222 — Lu AG09222 will be administered per schedule specified in the arm description.
  Arms: Lu AG09222 High Dose; Lu AG09222 Low Dose
Drug: Placebo — Placebo matching to Lu AG09222 will be administered per schedule specified in the arm description.
  Arms: Placebo

SUMMARY:
The main goal of this trial is to learn more about the safety of repeated dosing with Lu AG09222. The trial doctors will keep track of the participant's overall health by asking them how they are and by analyzing blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) ≥18.0 and ≤30 kilograms (kg)/square meter (m^2) at the screening visit.
* The participant has a clinical history of grass pollen allergic rhinitis of at least 2 years' duration as diagnosed by a physician.
* The participant has a positive specific immunoglobulin E (IgE) (defined as ≥class 2, ≥0.70 kilounits [kU]/liter [L]) against Phleum pratense at screening.
* The participant has a positive skin prick test with a wheal size ≥3 mm to Phleum pratense at screening.
* The participant is, in the opinion of the investigator, generally healthy based on medical history (despite the allergic rhinitis), a physical examination, vital signs, an electrocardiogram (ECG), and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The participant has received sublingual or subcutaneous immunotherapy with Phleum pratense within the last 5 years.
* The participant is receiving ongoing treatment with any allergy immunotherapy product.
* The participant has a clinically relevant history of symptomatic (seasonal or perennial) allergy caused by an allergen source overlapping with the allergen challenge period.
* The participant has taken disallowed medication or received a COVID-19 vaccination within the protocol-specified amount of time before Day 1.
* The participant has a relevant history of systemic allergic reaction, for example anaphylaxis with cardiorespiratory symptoms, generalized urticaria, or severe facial angioedema, which in the opinion of the investigator may constitute an increased safety concern.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Baseline (Day 1) up to Week 20

SECONDARY OUTCOMES:
Area Under the Serum Concentration-Time Curve in the Last Dosing Interval (AUC0-τ) of Lu AG09222 | Up to 96 hours post last dose on Days 57 to 61; and on Days 64, 71, 78, and 84
Maximum Observed Concentration (Cmax) of Lu AG09222 | Predose on Days 1 and 57; up to 96 hours post last dose on Days 57 to 61; and on Days 64, 71, 78, and 84
Time to Maximum Observed Concentration (Tmax) of Lu AG09222 | Predose on Days 1 and 57; up to 96 hours post last dose on Days 57 to 61; and on Days 64, 71, 78, and 84
Apparent Elimination Half-Life of Lu AG09222 | Predose on Days 1 and 57; up to 96 hours post last dose on Days 57 to 61; and on Days 64, 71, 78, and 84
Change from Baseline to Week 8 in Wheal-Reaction Area at 20 and 120 Minutes After Allergen Challenge | Baseline, Week 8
Change from Baseline to Week 8 in Flare-Reaction Area at 20 and 120 Minutes After Allergen Challenge | Baseline, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (2):
- United Kingdom (2):
  - St Pancras Clinical Research, London
  - Medicines Evaluation Unit, Manchester